CLINICAL TRIAL: NCT05734638
Title: Self-Care and Blood Pressure for Women Caregivers of Black and African-Americans With Alzheimer's Disease or Other Memory Problems *
Brief Title: Stress and Blood Pressure Management for Caregivers
Acronym: Stress/HTN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Kathy D. Wright, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2022B0064
Record Dates: First submitted 2022-11-10; First posted 2023-02-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Stress, Psychological
Keywords: Dementia Caregivers
MeSH Terms: conditions — Hypertension; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Randomized control trial of behavioral intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MIM-DASH (Experimental): A trained MIM provider (layperson) and a registered dietitian will deliver the MIM DASH group intervention in eight 1-hour (30 minutes MIM and 30 minutes DASH) sessions via telehealth (video and telephone access).
  Interventions: Behavioral: MIM-DASH
- MIM Only (Experimental): The MIM-only intervention group will receive the MIM education only in eight weekly sessions of 30 minutes each. To maintain equipoise among the intervention groups, this group will also have 30 minutes of "social time" to interact with the trainer and peers.
  Interventions: Behavioral: MIM Only
- DASH Only (Experimental): The DASH-only group will receive the DASH education only in eight weekly sessions of 30 minutes each. This group will also have 30 minutes of "social time" to interact with the trainer and peers, will receive their education from a different interventionist (also a registered dietician) and receive two coaching calls per month for 3 months, in this case focused on healthy eating DASH principles.
  Interventions: Behavioral: DASH Only

INTERVENTIONS:
Behavioral: MIM-DASH — Randomized participants will receive the MIM DASH, MIM or DASH intervention in eight weekly, 1-hour group sessions via telehealth (video and telephone access). Participants will receive session materials such as PowerPoint presentations so they can follow along by phone or videoconferencing. After completion of the eight weekly sessions, the participants will receive one follow-up call every other week for 8 weeks. The 3- and 6-month data will be collected as listed in the study AIMs. A manual of operations will detail all procedures related to the protocol, including participant recruitment, data collection, database usage, and database management.
  Arms: MIM-DASH
Behavioral: MIM Only — The MIM-only intervention group will receive the MIM education only in eight weekly sessions of 30 minutes each. To maintain equipoise among the intervention groups, this group will also have 30 minutes of "social time" to interact with the trainer and peers. To avoid cross contamination, the interventionist will not also deliver the intervention to the MIM DASH group. Each participant will have access to the digital meditations with mindfulness practice recordings as well as a weekly diary to document study activities. Participants will be instructed to perform mindfulness meditations at least five times a week and record the time in their diary. After completion of the eight weekly sessions, these participants will receive six coaching calls (two per month for 3 months) focused on mindfulness practice.
  Arms: MIM Only
Behavioral: DASH Only — The DASH-only group will receive the DASH education only in eight weekly sessions of 30 minutes each. This group will also have 30 minutes of "social time" to interact with the trainer and peers, will receive their education from a different interventionist (also a registered dietician) and receive two coaching calls per month for 3 months, in this case focused on healthy eating DASH principles.
  Arms: DASH Only

SUMMARY:
Due to health and wealth disparities, no demographic group is more at risk than African American women for the double jeopardy of stress from caregiving for persons living with dementia (PLWD) and stress associated with hypertension (HTN). This double jeopardy puts those they care for in jeopardy as well: Reduced quality of life and longevity, disability, cognitive decline, and stroke associated with HTN1 impede caregiving activities and resultant health and well-being for persons living with Alzheimer's disease and related dementias (ADRD). Although successful multi-component interventions have addressed ADRD caregiver stress (REACH II) and the Savvy Caregiver program, to our knowledge there are no interventions that target the complexity of chronic caregiving stress and HTN self-care for African American women caregivers of persons living with ADRD.

This project will test two interventions for their effectiveness in improving outcomes for the target group: Mindfulness in Motion (MIM) and the Dietary Approaches to Stop Hypertension (DASH). MIM includes mindful awareness and movement from a seated position, breathing exercises, healthy sleep, and guided mindfulness meditation. The DASH component will be tailored for Black Americans. It uses a critical thinking approach that involves problem solving, participant-centered goal setting, health coaching, reflection, and development of self-efficacy (confidence) to promote physical activity and healthy eating. Solid empirical evidence demonstrates its effectiveness in reducing blood pressure among mixed-race samples.

DETAILED DESCRIPTION:
Our long-term goal is to develop effective interventions to reduce cardiovascular health disparities and improve health outcomes among African American women. Given this gap in knowledge (i.e., interventions targeting caregiving stress and hypertension self-care), our Stage I pilot study focuses on a) caregiver stress and b) self-care for hypertension, the most prevalent chronic condition among African American women caregivers of PLWD. We know lifestyle changes are effective in managing HTN, but they will not make a difference in controlling hypertension if individuals do not engage in these health behaviors. Unfortunately, African American women are less likely to engage in self-care (such as diet and exercise behaviors) if they believe their hypertension is caused by stress. Indeed, our past research demonstrates that stressful interpersonal communication problems, blood pressure knowledge deficits, and complex diet information all interfered with older African American women's blood pressure self-care. Thus, we investigate the hypothesis that by addressing stress reactivity/stress resilience as the underlying mechanism to facilitate behavioral change, the intervention will be successful in enhancing HTN self-care.

A small-scale, Stage I, three-group randomized controlled trial (RCT) will investigate the feasibility of MIM plus DASH to improve blood pressure self-care in African American caregivers, as compared to MIM only or DASH only. Each intervention will be delivered in eight weekly 1-hour group sessions via telehealth.

To our knowledge, this is the first study that systematically a) examines impact on self-care behaviors and b) employs one of the Science of Behavioral Change key mechanisms underlying successful change in health behaviors-stress reactivity/stress resilience among a large, underrepresented demographic group. PI Wright will recruit 90 women with hypertension who are caring for persons living with ADRD, 30 per group (MIM DASH, MIM only, or DASH only). We will collect data at baseline, 3-months, and 6-months. The interprofessional team pursuing this project has worked together for 3 years. Our aims will be as follows:

AIM 1. Determine the feasibility of MIM DASH, MIM, and DASH for African American women caregivers of family/friends living with dementia. Hypothesis: African American women caregivers with hypertension will participate in the MIM DASH as well as the active control groups (MIM or DASH).

Aim 2. Examine pilot efficacy of the MIM DASH intervention to improve stress and self-care as compared to active control groups (MIM or DASH). Hypothesis: Stress will be reduced and self-care will be improved in the MIM DASH group as compared to active control groups (MIM or DASH).

AIM 3. Examine the pilot efficacy of the combination of MIM plus DASH for improvement of systolic blood pressure (SBP) as compared to active control groups (MIM or DASH). Hypothesis: Relative to baseline assessment, the MIM DASH group will exhibit lower SBP at 3 and 6 months as compared to active control groups (MIM or DASH).

ELIGIBILITY:
Inclusion criteria are (1) diagnosis of HTN treated with an antihypertensive medication; (2) age 40 and older (3) a caregiver rating of the PLWD of 2 or greater on the Alzheimer's Dementia-8 scale;50 (4) providing unpaid care to a PLWD at least 10 hours per week or assisting with at least one instrumental activity of daily living (5) self-identifies as Black/African American; (6) English speaking; and (7) has access to a telecommunications device such as the internet via desktop, laptop/tablet, smartphone, or telephone.

Exclusion criteria are (1) diagnosis of resistant HTN (blood pressure that remains above goal despite concurrent use of a diuretic/water pill and at least two other antihypertensive agents of different classes); or (2) active participation in mindfulness/yoga program.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | Baseline, 3 months, 6 months
  Systolic and Diastolic blood pressure measured with automatic blood pressure cuff. Results outside of the normal range (90/60 to 120/80 mmHg), both higher and lower are considered undesirable.

SECONDARY OUTCOMES:
Hair Cortisol | Baseline, 6 months
  Hair cortisol (HC) will be used as a proxy for chronic stress. Approximately 25-75 mg of hair will be cut from the posterior vertex region of the scalp as close to the scalp as possible. Participants will be surveyed on corticosteroid use as these medications may suppress cortisol levels, and on their hair care practices, such as frequency of washing, chemical treatments and hair product use. Hair Cortisol levels are expressed in hair as pg/mg and generally logged due to skewed distributions as needed. Higher levels of cortisol indicated higher levels of chronic stress and a less desirable outcome.
Block food frequency questionnaire | Baseline, 3 months, 6 months
  Block Food Frequency Questionnaire (includes physical activity) is a validated measure with a food and beverage list that includes 127 items, plus supplementary questions to allow for the adjustment of fat, protein, carbohydrate, sugar, and whole grain content. The questionnaire ascertains the frequency with which each food or beverage was usually consumed, and offers nine continuous responses ranging from "never" to "every day" for most foods. The DASH Index that is calculated using data from the Block Food Frequency Questionnaire uses a quintile system to score foods related to the DASH diet. All of the components are equally weighted. Intake of vegetables, fruits (including fruit juice), nuts and legumes, whole grains were scored from 1 (lowest quintile) to 5 (highest quintile). The overall DASH component scores range from 8 to 40. With higher scores indicating healthier diets
Daily inventory of stressful events | Baseline, 3 months, 6 months
  The instrument is a semi-structured survey in which participants report whether any stressful events had occurred within the past 24 hours. This instrument yields several variables for each reported stressor including: (a) content classification of the stressor for example, work overload, argument over housework, or traffic problem); (b) subjective severity of stressors; (c) primary appraisals (areas of life that were at risk because of the stressor); and (d) perceived control of the situation." Scores range from 0 to 27. Higher scores indicate more stressful events.
Perceived stress scale (caregiver stress) | Baseline, 3 months, 6 months
  The Perceived Stress Scale has 10-items one a Likert scale with a reference range of 0-30 regarding stress over the past month. Values are: 0 - Never, 1 - Almost Never, 2 - Sometimes, 3 - Fairly Often, 4 - Very Often The investigators will sum 10 items to create a composite score, ranging from 0 to 40.
  The higher score, the higher levels of perceived stress.
Depression Anxiety Stress Symptom Scale (DASS-21) | Baseline, 3 months, 6 months
  Assess psychological comorbidity of the caregiver and health status of the person living with ADRD. Contains 21 items to evaluate mild, moderate, or severe depression, anxiety, and stress (α =0.79). Scores range from 0-37 with higher scores indicating more symptoms.
Revised Memory and Behavior Checklist | Baseline, 3 months, 6 months
  Assess psychological comorbidity of the caregiver and health status of the person living with ADRD. 32-item check-list that assess activities of daily living and problem behaviors in people living with ADRD. Scores range from 0-96 with higher indicating more behavioral problems in the care recipient
Credibility Scale | 3 months
  The Credibility Scale (α = 0.86) measures attitudes towards the treatment condition and the participants' expectation of benefit once the treatment has been explained. The scale consists of 5 questions rated on a 0 (not at all confident) to 10 (very confident). Higher scores, up to 45, will indicate greater credibility of the treatment condition.
Acceptability Scale | 3 months
  Treatment-specific preference ratings (pre- and post-intervention).The participants will complete the Acceptability of Participant Preferences 13-item Likert-type survey ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate that participants find the intervention more acceptable.
Krousel-Wood Medication Adherence Scale | Baseline, 3 months, 6 months
  The 4-Item scale captures four domains of adherence behavior. Scores range from 0 to 4 with a score of 1 or greater indicating lower adherence.
Patient Health Questionnaire (PHQ-9) | Baseline, 3 months, 6 months
  The PHQ-9 is a 9-item measure of depression and each item is scored on a scale of 0-3. The total ranges from 0-27 (scores of 5-9 are mild depression, 10-14 are moderate depression, 15-19 are moderately severe depression, ansd 20 and above are severe depression.)
Generalized Anxiety Disorder Scale (GAD-7) | Baseline, 3 months, 6 months
  GAD-7 is a 7-item self-admiistered tool used to measure generalized anxiety. Each item is scored on a scale of 0-3, with the total ranging from 0-21 points. Scores of 5-9 indicate mild anxiety, 10-14 indicate moderate anxiety, and 15 and more indicate severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Wright, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be disseminated using multiple strategies, such as making our results available to the NIH ClinicalTrials.gov website, transmitting them to the aging research community through peer-reviewed journals, and giving presentations of the results of the study at national and international scientific meetings. Additionally, presentations will be given to the local African American community to churches, Alzheimer's disease support groups, and beauty salons.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available 01/01/2027 until 0101/2027
Access Criteria: To access data, inquires will go to Kathy Wright, PhD, RN at wright.2104@osu.edu

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT05734638/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT05734638/ICF_001.pdf